CLINICAL TRIAL: NCT00514735
Title: Tailored Treatment of Permanent Atrial Fibrillation - TTOP-AF
Brief Title: Tailored Treatment of Permanent Atrial Fibrillation
Acronym: TTOP-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFI-30
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Results first posted 2012-05-09 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ablation Management
  Interventions: Procedure: Medtronic Cardiac Ablation System
- 2 (Active Comparator): Medical Management
  Interventions: Drug: Class I or III Antiarrhythmic Medications

INTERVENTIONS:
Procedure: Medtronic Cardiac Ablation System — Arm 1 (Ablation Management): Ablation procedures using investigational catheters in left atrium. Cardioversion could be used to restore sinus rhythm if needed.
  Arms: 1
Drug: Class I or III Antiarrhythmic Medications — Arm 2 (Medical Management): Class I or III antiarrhythmic drugs. Changes in dosing, antiarrhythmic drugs or combinations of antiarrhythmic drugs were allowed. Direct current cardioversions were also allowed at the discretion of the investigator.
  Arms: 2

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of the Medtronic Cardiac Ablation System compared to medical therapy in the persistent and long-standing persistent atrial fibrillation population.

ELIGIBILITY:
INCLUSION CRITERIA:

* History of symptomatic, continuous atrial fibrillation defined as: Continuous atrial fibrillation lasting greater than 1 year but less than 4 years or nonself-terminating atrial fibrillation, lasting greater than 7 days but no more than 1 year, with at least one failed direct current cardioversion. A failed cardioversion was defined as an unsuccessful cardioversion or one in which normal sinus rhythm was established but not maintained beyond 7 days.
* Atrial fibrillation symptoms included the following: palpitations, fatigue,exertional dyspnea, exercise intolerance
* Age between 18 and 70 years
* Failure of at least one Class I or III rhythm control drug
* Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study.

EXCLUSION CRITERIA:

* Structural heart disease of clinical significance including:

  * Previous cardiac surgery (excluding coronary artery bypass graft and mitral valve repair)
  * Symptoms of congestive heart failure including, but not limited to, New York Heart Association (NYHA) Class III or IV congestive heart failure and/or documented ejection fraction <40% measured by acceptable cardiac testing
  * Left atrial diameter >55 mm
  * Moderate to severe mitral or aortic valvular heart disease
  * Stable/unstable angina or ongoing myocardial ischemia
  * Myocardial infarction (MI) within 3 months of enrollment
  * Congenital heart disease (not including atrial septal defect or patent foramen ovale without a right to left shunt) where the underlying abnormality increases the risk of an ablative procedure
  * Prior atrial septal defect of patent foramen ovale closure with a device using a percutaneous approach
  * Hypertrophic cardiomyopathy (left ventricular septal wall thickness >1.5 cm)
  * Pulmonary hypertension (mean or systolic pulmonary artery pressure >50 mm Hg on Doppler echo)
* Any prior ablation for atrial fibrillation
* Enrollment in any other ongoing arrhythmia study
* Any ventricular tachyarrhythmia currently being treated where the arrhythmia or the management may interfere with this study
* Active infection or sepsis
* Any history of cerebral vascular disease including stroke or transient ischemic attacks
* Pregnancy or lactation
* Left atrial thrombus at the time of ablation
* Untreatable allergy to contrast media
* Any diagnosis of atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiovascular causes
* History of blood clotting (bleeding or thrombotic) abnormalities
* Known sensitivities to heparin or warfarin
* Severe chronic obstructive pulmonary disease (defined as forced expiratory volume 1 (FEV1) <1)
* Severe co-morbidity or poor general physical/mental health that, in the opinion of the investigator, will not allow the subject to be a good study candidate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (23):
  - Arizona Arrhythmia Research Center, Scottsdale, Arizona
  - UCLA Cardiac Arrhythmia Center, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - Iowa Heart Center, Des Moines, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Massachusetts General Hospital Cardiac Arrhythmia, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health Research Department, Grand Rapids, Michigan
  - University of Rochester, Rochester, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Consultants in Cardiovascular Diseases, Erie, Pennsylvania
  - Austin Heart, Austin, Texas
  - Texas Heart Institute at St. Luke's Episcopal, Houston, Texas
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands

REFERENCES:
- [Background] Fuster V, Ryden LE, Asinger RW, Cannom DS, Crijns HJ, Frye RL, Halperin JL, Kay GN, Klein WW, Levy S, McNamara RL, Prystowsky EN, Wann LS, Wyse DG, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO, Smith SC, Klein WW, Alonso-Garcia A, Blomstrom-Lundqvist C, De Backer G, Flather M, Hradec J, Oto A, Parkhomenko A, Silber S, Torbicki A; American College of Cardiology/American Heart Association/European Society of Cardiology Board. ACC/AHA/ESC guidelines for the management of patients with atrial fibrillation: executive summary. A Report of the American College of Cardiology/ American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines and Policy Conferences (Committee to Develop Guidelines for the Management of Patients With Atrial Fibrillation): developed in Collaboration With the North American Society of Pacing and Electrophysiology. J Am Coll Cardiol. 2001 Oct;38(4):1231-66. doi: 10.1016/s0735-1097(01)01587-x. No abstract available. PMID 11583910
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Halperin JL, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 Guidelines for the Management of Patients with Atrial Fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006 Aug 15;114(7):e257-354. doi: 10.1161/CIRCULATIONAHA.106.177292. No abstract available. PMID 16908781
- [Background] Benussi S, Nascimbene S, Calori G, Denti P, Ziskind Z, Kassem S, La Canna G, Pappone C, Alfieri O. Surgical ablation of atrial fibrillation with a novel bipolar radiofrequency device. J Thorac Cardiovasc Surg. 2005 Aug;130(2):491-7. doi: 10.1016/j.jtcvs.2005.01.009. PMID 16077418
- [Background] Dill T, Neumann T, Ekinci O, Breidenbach C, John A, Erdogan A, Bachmann G, Hamm CW, Pitschner HF. Pulmonary vein diameter reduction after radiofrequency catheter ablation for paroxysmal atrial fibrillation evaluated by contrast-enhanced three-dimensional magnetic resonance imaging. Circulation. 2003 Feb 18;107(6):845-50. doi: 10.1161/01.cir.0000048146.81336.1d. PMID 12591754
- [Background] Dong J, Vasamreddy CR, Jayam V, Dalal D, Dickfeld T, Eldadah Z, Meininger G, Halperin HR, Berger R, Bluemke DA, Calkins H. Incidence and predictors of pulmonary vein stenosis following catheter ablation of atrial fibrillation using the anatomic pulmonary vein ablation approach: results from paired magnetic resonance imaging. J Cardiovasc Electrophysiol. 2005 Aug;16(8):845-52. doi: 10.1111/j.1540-8167.2005.40680.x. PMID 16101625
- [Background] Food and Drug Administration Guidance for Industry and FDA Staff: Clinical Study Designs for Percutaneous Catheter Ablation for Treatment of Atrial Fibrillation, January 9, 2004.
- [Background] Abreu Filho CA, Lisboa LA, Dallan LA, Spina GS, Grinberg M, Scanavacca M, Sosa EA, Ramires JA, Oliveira SA. Effectiveness of the maze procedure using cooled-tip radiofrequency ablation in patients with permanent atrial fibrillation and rheumatic mitral valve disease. Circulation. 2005 Aug 30;112(9 Suppl):I20-5. doi: 10.1161/CIRCULATIONAHA.104.526301. PMID 16159816
- [Background] Fisher JD, Spinelli MA, Mookherjee D, Krumerman AK, Palma EC. Atrial fibrillation ablation: reaching the mainstream. Pacing Clin Electrophysiol. 2006 May;29(5):523-37. doi: 10.1111/j.1540-8159.2006.00388.x. PMID 16689850
- [Background] Gajewski J, Singer RB. Mortality in an insured population with atrial fibrillation. JAMA. 1981 Apr 17;245(15):1540-4. PMID 7206163
- [Background] de Lima GG, Kalil RA, Leiria TL, Hatem DM, Kruse CL, Abrahao R, Sant'anna JR, Prates PR, Nesralla IA. Randomized study of surgery for patients with permanent atrial fibrillation as a result of mitral valve disease. Ann Thorac Surg. 2004 Jun;77(6):2089-94; discussion 2094-5. doi: 10.1016/j.athoracsur.2003.11.018. PMID 15172273
- [Background] Hindricks G, Piorkowski C, Tanner H, Kobza R, Gerds-Li JH, Carbucicchio C, Kottkamp H. Perception of atrial fibrillation before and after radiofrequency catheter ablation: relevance of asymptomatic arrhythmia recurrence. Circulation. 2005 Jul 19;112(3):307-13. doi: 10.1161/CIRCULATIONAHA.104.518837. Epub 2005 Jul 11. PMID 16009793
- [Background] Hornero F, Rodriguez I, Bueno M, Buendia J, Dalmau MJ, Canovas S, Gil O, Garcia R, Montero JA. Surgical ablation of permanent atrial fibrillation by means of maze radiofrequency: mid-term results. J Card Surg. 2004 Sep-Oct;19(5):383-8. doi: 10.1111/j.0886-0440.2004.04077.x. PMID 15383047
- [Background] Kerr CR, Humphries KH, Talajic M, Klein GJ, Connolly SJ, Green M, Boone J, Sheldon R, Dorian P, Newman D. Progression to chronic atrial fibrillation after the initial diagnosis of paroxysmal atrial fibrillation: results from the Canadian Registry of Atrial Fibrillation. Am Heart J. 2005 Mar;149(3):489-96. doi: 10.1016/j.ahj.2004.09.053. PMID 15864238
- [Background] Marrouche NF, Martin DO, Wazni O, Gillinov AM, Klein A, Bhargava M, Saad E, Bash D, Yamada H, Jaber W, Schweikert R, Tchou P, Abdul-Karim A, Saliba W, Natale A. Phased-array intracardiac echocardiography monitoring during pulmonary vein isolation in patients with atrial fibrillation: impact on outcome and complications. Circulation. 2003 Jun 3;107(21):2710-6. doi: 10.1161/01.CIR.0000070541.83326.15. Epub 2003 May 19. PMID 12756153
- [Background] Nademanee K, McKenzie J, Kosar E, Schwab M, Sunsaneewitayakul B, Vasavakul T, Khunnawat C, Ngarmukos T. A new approach for catheter ablation of atrial fibrillation: mapping of the electrophysiologic substrate. J Am Coll Cardiol. 2004 Jun 2;43(11):2044-53. doi: 10.1016/j.jacc.2003.12.054. PMID 15172410
- [Background] Oral H, Pappone C, Chugh A, Good E, Bogun F, Pelosi F Jr, Bates ER, Lehmann MH, Vicedomini G, Augello G, Agricola E, Sala S, Santinelli V, Morady F. Circumferential pulmonary-vein ablation for chronic atrial fibrillation. N Engl J Med. 2006 Mar 2;354(9):934-41. doi: 10.1056/NEJMoa050955. PMID 16510747
- [Background] Packer DL, Asirvatham S, Munger TM. Progress in nonpharmacologic therapy of atrial fibrillation. J Cardiovasc Electrophysiol. 2003 Dec;14(12 Suppl):S296-309. doi: 10.1046/j.1540-8167.2003.90403.x. No abstract available. PMID 15005218
- [Background] Pappone C, Rosanio S, Augello G, Gallus G, Vicedomini G, Mazzone P, Gulletta S, Gugliotta F, Pappone A, Santinelli V, Tortoriello V, Sala S, Zangrillo A, Crescenzi G, Benussi S, Alfieri O. Mortality, morbidity, and quality of life after circumferential pulmonary vein ablation for atrial fibrillation: outcomes from a controlled nonrandomized long-term study. J Am Coll Cardiol. 2003 Jul 16;42(2):185-97. doi: 10.1016/s0735-1097(03)00577-1. PMID 12875749
- [Background] PMA P020025 - Summary of Safety and Effectiveness Data: Boston Scientific Corporation Blazer II XP™ Cardiac Ablation Catheter, August 25, 2003.
- [Background] PMA P030031 - Summary of Safety and Effectiveness Data: Biosense Webster Navistar™/Celsius™ThermoCool® Diagnostic/Ablation Deflectable Tip Catheters, November 5, 2004.
- [Background] PMA P040042 - Summary of Safety and Effectiveness Data: Irvine Biomedical, Inc. IBI Therapy™ Dual 8™ Ablation Catheter, November 18, 2005.
- [Background] Saad EB, Cole CR, Marrouche NF, Dresing TJ, Perez-Lugones A, Saliba WI, Schweikert RA, Klein A, Rodriguez L, Grimm R, Tchou P, Natale A. Use of intracardiac echocardiography for prediction of chronic pulmonary vein stenosis after ablation of atrial fibrillation. J Cardiovasc Electrophysiol. 2002 Oct;13(10):986-9. doi: 10.1046/j.1540-8167.2002.00986.x. PMID 12435183
- [Background] Saad EB, Rossillo A, Saad CP, Martin DO, Bhargava M, Erciyes D, Bash D, Williams-Andrews M, Beheiry S, Marrouche NF, Adams J, Pisano E, Fanelli R, Potenza D, Raviele A, Bonso A, Themistoclakis S, Brachmann J, Saliba WI, Schweikert RA, Natale A. Pulmonary vein stenosis after radiofrequency ablation of atrial fibrillation: functional characterization, evolution, and influence of the ablation strategy. Circulation. 2003 Dec 23;108(25):3102-7. doi: 10.1161/01.CIR.0000104569.96907.7F. Epub 2003 Nov 17. PMID 14623799
- [Background] Scardi S, Mazzone C, Pandullo C, Goldstein D, Poletti A, Humar F. Lone atrial fibrillation: prognostic differences between paroxysmal and chronic forms after 10 years of follow-up. Am Heart J. 1999 Apr;137(4 Pt 1):686-91. doi: 10.1016/s0002-8703(99)70224-3. PMID 10097231
- [Background] Vasamreddy CR, Dalal D, Dong J, Cheng A, Spragg D, Lamiy SZ, Meininger G, Henrikson CA, Marine JE, Berger R, Calkins H. Symptomatic and asymptomatic atrial fibrillation in patients undergoing radiofrequency catheter ablation. J Cardiovasc Electrophysiol. 2006 Feb;17(2):134-9. doi: 10.1111/j.1540-8167.2006.00359.x. PMID 16533249
- [Background] Vasamreddy CR, Dalal D, Eldadah Z, Dickfeld T, Jayam VK, Henrickson C, Meininger G, Dong J, Lickfett L, Berger R, Calkins H. Safety and efficacy of circumferential pulmonary vein catheter ablation of atrial fibrillation. Heart Rhythm. 2005 Jan;2(1):42-8. doi: 10.1016/j.hrthm.2004.10.027. PMID 15851264
- [Background] Wazni OM, Marrouche NF, Martin DO, Verma A, Bhargava M, Saliba W, Bash D, Schweikert R, Brachmann J, Gunther J, Gutleben K, Pisano E, Potenza D, Fanelli R, Raviele A, Themistoclakis S, Rossillo A, Bonso A, Natale A. Radiofrequency ablation vs antiarrhythmic drugs as first-line treatment of symptomatic atrial fibrillation: a randomized trial. JAMA. 2005 Jun 1;293(21):2634-40. doi: 10.1001/jama.293.21.2634. PMID 15928285
- [Background] Chen YJ, Chen SA, Tai CT, Wen ZC, Feng AN, Ding YA, Chang MS. Role of atrial electrophysiology and autonomic nervous system in patients with supraventricular tachycardia and paroxysmal atrial fibrillation. J Am Coll Cardiol. 1998 Sep;32(3):732-8. doi: 10.1016/s0735-1097(98)00305-2. PMID 9741520
- [Background] Haissaguerre M, Sanders P, Hocini M, Hsu LF, Shah DC, Scavee C, Takahashi Y, Rotter M, Pasquie JL, Garrigue S, Clementy J, Jais P. Changes in atrial fibrillation cycle length and inducibility during catheter ablation and their relation to outcome. Circulation. 2004 Jun 22;109(24):3007-13. doi: 10.1161/01.CIR.0000130645.95357.97. Epub 2004 Jun 7. PMID 15184286
- [Background] Sanders P, Nalliah CJ, Dubois R, Takahashi Y, Hocini M, Rotter M, Rostock T, Sacher F, Hsu LF, Jonsson A, O'Neill MD, Jais P, Haissaguerre M. Frequency mapping of the pulmonary veins in paroxysmal versus permanent atrial fibrillation. J Cardiovasc Electrophysiol. 2006 Sep;17(9):965-72. doi: 10.1111/j.1540-8167.2006.00546.x. PMID 16948740
- [Background] Jais P, Hocini M, Sanders P, Hsu LF, Takahashi Y, Rotter M, Rostock T, Sacher F, Clementy J, Haissaguerre M. Long-term evaluation of atrial fibrillation ablation guided by noninducibility. Heart Rhythm. 2006 Feb;3(2):140-5. doi: 10.1016/j.hrthm.2005.11.012. PMID 16443526
- [Background] Earley MJ, Abrams DJ, Staniforth AD, Sporton SC, Schilling RJ. Catheter ablation of permanent atrial fibrillation: medium term results. Heart. 2006 Feb;92(2):233-8. doi: 10.1136/hrt.2005.066969. Epub 2005 Aug 23. PMID 16118239
- [Background] Nilsson B, Chen X, Pehrson S, Kober L, Hilden J, Svendsen JH. Recurrence of pulmonary vein conduction and atrial fibrillation after pulmonary vein isolation for atrial fibrillation: a randomized trial of the ostial versus the extraostial ablation strategy. Am Heart J. 2006 Sep;152(3):537.e1-8. doi: 10.1016/j.ahj.2006.05.029. PMID 16923426
- [Background] Rotter M, Takahashi Y, Sanders P, Haissaguerre M, Jais P, Hsu LF, Sacher F, Pasquie JL, Clementy J, Hocini M. Reduction of fluoroscopy exposure and procedure duration during ablation of atrial fibrillation using a novel anatomical navigation system. Eur Heart J. 2005 Jul;26(14):1415-21. doi: 10.1093/eurheartj/ehi172. Epub 2005 Mar 1. PMID 15741228
- See also: Company website — http://www.ablationfrontiers.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on November 28, 2007. The very last ablation procedure was a retreatment ablation procedure for a Medical Management Crossover subject that occurred on May 7, 2010 with the final follow-up on November 1, 2010.
Pre-assignment Details: 32 subjects signed Informed Consent forms but withdrew from the study prior to randomization.
  * 24 failed to meet inclusion/exclusion criteria
  * 6 elected to withdraw
  * 1 subject was withdrawn by the Sponsor after being consented.
  * 1 subject was withdrawn as screening was incomplete prior to closing enrollment for the study
Groups:
- Ablation Management: Pre- and post- procedure anticoagulation was managed according to the preference of the investigator. Left atrial access was obtained by a single transseptal puncture. No ablations were to occur until the activated clotting time reached 300 seconds, which was to be maintained for the duration of the ablation. During the index ablation procedure, investigators were required to use all 3 investigational catheters. Cardioversion could be used to restore sinus rhythm if needed. If there was a recurrence of atrial fibrillation, a repeat ablation procedure could be performed any time during the follow-up period. With a retreatment, the follow-up clock was restarted. Subjects were seen pre-discharge and at in-clinic follow-up visits at 1, 3, and 6 months.
- Medical Management: Medical Management subjects were prescribed Class I or III antiarrhythmic drugs. Changes in dosing, antiarrhythmic drugs or combinations of antiarrhythmic drugs were allowed. Direct current (DC) cardioversions were also allowed at the discretion of the investigator. Anticoagulation was to be maintained at an International Normalized Ratio greater than 2. Subjects were seen at in-clinic follow-up visits at 1, 3, and 6 months. Subjects who demonstrated chronic treatment failure while under drug therapy could cross over, and receive an ablation as early as 4 months post randomization.
Period: Overall Study
Arm/Group | Ablation Management | Medical Management
Started | 138 | 72
Completed | 124 | 66
Not Completed | 14 | 6
Not completed — Withdrawal by Subject | 13 | 5
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ablation Management | Medical Management | Total
Number analyzed (Participants) | 138 | 72 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 43 | 136
  >=65 years | 45 | 29 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (8.3) | 60.7 (8.9) | 60.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 115 | 60 | 175
Region of Enrollment [Number; unit: participants]
  United States | 126 | 65 | 191
  Netherlands | 12 | 7 | 19
Number of DC cardioversions in past 4 years [Mean (Standard Deviation); unit: cardioversions] — Number of DC cardioversions in past 4 years per subject
  cardioversions | 2.0 (1.1) | 2.4 (3.5) | 2.1 (2.2)
Number of previously failed AADs per subject [Mean (Standard Deviation); unit: antiarrhythmic drugs] | 1.4 (0.6) | 1.1 (0.4) | 1.3 (0.6)
Left Atrial Diameter [Mean (Standard Deviation); unit: centimeters] | 4.5 (0.5) | 4.6 (0.5) | 4.6 (0.5)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percent] | 54.7 (7.1) | 54.9 (6.7) | 54.7 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Chronic Effectiveness
Description: The chronic efficacy endpoint was a treatment success/failure measure for each subject computed at 6 months. Treatment success included:
  1. A 90% reduction in clinically significant atrial fibrillation from baseline to the 6 month time point based on a Holter recording. Clinically significant atrial fibrillation was defined as sustained atrial fibrillation lasting more than 10 minutes.
  2. The subject was off all antiarrhythmic drugs at 6 months (Ablation Management arm only)
  3. The Investigator judged all procedures to be acutely successful (Ablation Management arm only).
Time Frame: 6 months
Population: An Intention to Treat (ITT) analysis was performed in which all data was analyzed according to the subject's assigned randomization group. The primary missing value imputation technique for all primary endpoint analyses was the passive method of imputation.
Measure: Number; unit: percentage of participants with success
Arm/Group | Ablation Management | Medical Management
Number analyzed (Participants) | 138 | 72
percentage of participants with success | 56 | 26
Statistical Analysis 1: Comparison: Ablation Management vs Medical Management; H0: Pa ≤ Pm Ha: Pa > Pm where Pa is the proportion of successfully treated subjects in the ablation management arm and Pm is the proportion of successfully treated subjects in the optimal medical management/drug therapy arm; Test type: Superiority or Other; p < 0.0001, Chi-squared — In order to maintain the overall level of significance at the α=0.025 level after a planned interim analysis using α=0.003, this test will actually be performed using an adjusted α=0.0245 at the completion of the study

2. Primary Outcome: Acute Safety
Description: The primary endpoint for acute safety was a success/failure variable calculated for each subject in Ablation Management at the 7 day post-procedure time point. Any subject with at least one adverse event adjudicated by the Data Safety Monitoring Board as both serious and either probably or definitely procedure and/or device-related occurring within 7 days of the ablation procedure was considered an acute safety failure, regardless of whether the event occurred following the index or retreatment ablation procedure.
Time Frame: 7 days
Population: An Intention to Treat (ITT) analysis was performed in which all data was analyzed according to the subject's assigned randomization group.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ablation Management
Number analyzed (Participants) | 138
percentage of participants | 12.3 [7.3 to 19.0]
Statistical Analysis 1: Comparison: Ablation Management; H0: Pa ≥ 0.16 Ha: Pa < 0.16 where Pa is the proportion of acute safety failures in the ablation management arm; Test type: Superiority or Other; p = 0.1427, Fisher Exact — An exact, one-sample binomial test was conducted at a one-sided α=0.025 level of significance

3. Primary Outcome: Chronic Safety
Description: The primary endpoint for chronic safety was a success/failure variable calculated for each subject at 6 months. Any subject that had at least one adverse event that met designated seriousness and relatedness criteria for the particular treatment group as adjudicated by the Data Safety Monitoring Board was considered a chronic safety failure. Adverse events in Ablation Management that were acute (≤7 days) were not included in the chronic safety primary endpoint. Given the disparity in the length of time at risk between treatment arms,the Chronic Safety endpoint was not statistically powered.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Medical Management: Medical Management subjects were prescribed Class I or III antiarrhythmic drugs. Changes in dosing, antiarrhythmic drugs or combinations of antiarrhythmic drugs were allowed. Direct current cardioversions were also allowed at the discretion of the investigator. Anticoagulation was to be maintained at an International Normalized Ratio greater than 2. Subjects were seen at in-clinic follow-up visits at 1, 3, and 6 months. Subjects who demonstrated chronic treatment failure while under drug therapy could cross over, and receive an ablation as early as 4 months post randomization.
Arm/Group | Ablation Management | Medical Management
Number analyzed (Participants) | 138 | 72
participants | 9 | 3
Statistical Analysis 1: Comparison: Ablation Management vs Medical Management; H0: Pa ≥ Pm + 0.06 Ha: Pa < Pm + 0.06 where Pa is the proportion of failed subjects in the ablation management arm and Pm is the proportion of failed subjects in the optimal medical management/drug therapy arm; Test type: Non-Inferiority or Equivalence — This objective was not statistically powered. The non-inferiority chronic safety margin was 0.06; p = 0.0033, t-test, 1 sided

4. Secondary Outcome: Acute Efficacy
Description: A treatment success/failure up to the conclusion of the procedure for each subject in Ablation Management. A subject was considered successfully treated if the following were true:
  * Medtronic ablation catheters were used to achieve procedure success.
  * All accessible pulmonary veins were isolated.
  * At least 50% reduction of complex fractionated atrial electrograms mapped and ablated with Medtronic ablation catheters.
  * Sinus rhythm was achieved upon leaving the electrophysiology lab (±cardioversion).
Time Frame: Procedure conclusion
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ablation Management
Number analyzed (Participants) | 138
percentage of participants | 92.8 [87 to 96]

5. Secondary Outcome: Improvement of Left Atrial Size at 6 Months Compared to Baseline.
Description: Left atrial diameter (LAD), as measured by transthoracic echocardiogram (TTE) looking at the longitudinal long axis at baseline and at the 6 month follow-up visit in both the Ablation and Medical Management arms.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Ablation Management | Medical Management
Number analyzed (Participants) | 138 | 72
centimeters
  Measurement at Baseline | 4.5 (0.53) | 4.6 (0.49)
  Measurement at 6 Months | 4.4 (0.67) | 4.6 (0.56)
Statistical Analysis 1: Comparison: Ablation Management vs Medical Management; H0: μa = μm Ha: μa ≠ μm where μa is the change of LAD from baseline to 6 month in Ablation Management arm, and μm is the change of LAD from baseline to 6 month in Medical Management arm; Test type: Superiority or Other; p = 0.35, ANOVA

6. Secondary Outcome: Improvement of Left Ventricular Ejection Fraction at 6 Months Compared to Baseline.
Description: Left ventricular ejection fraction (LVEF), as measured by transthoracic echocardiogram at baseline and 6 months in both the Ablation and Medical Management arms.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Ablation Management | Medical Management
Number analyzed (Participants) | 138 | 72
percent
  Measurement at Baseline | 54.7 (7.09) | 54.9 (6.73)
  Measurement at 6 Months | 58.3 (6.73) | 57.0 (6.06)
Statistical Analysis 1: Comparison: Ablation Management vs Medical Management; H0: μa = μm Ha: μa ≠ μm where μa is the change of LVEF from baseline to 6 month in Ablation Management arm, and μm is the change of LVEF from baseline to 6 month in Medical Management arm; Test type: Superiority or Other; p = 0.06, ANOVA

7. Secondary Outcome: Improvement in Atrial Fibrillation (AF) Symptom Severity Scores Over 6 Months Compared to Baseline.
Description: The severity of subject's atrial fibrillation related symptoms on a scale from 1 (no symptoms) to 5 (most severe). The symptoms included palpitations, fatigue, shortness of breath, lightheadedness or dizziness, and lack of energy during exertion or exercise. The scores were tabulated at the 1, 3 and 6 month follow-up visits. Scores could range from 5 to 25, indicating a spectrum of subject status from asymptomatic to severely symptomatic.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: AF Symptom Severity Score
Arm/Group | Ablation Management | Medical Management
Number analyzed (Participants) | 138 | 72
AF Symptom Severity Score
  Measurement at Baseline | 12.38 (4.21) | 12.72 (4.47)
  Measurement at 1 Month | 8.95 (3.58) | 9.90 (3.85)
  Measurement at 3 Months | 7.56 (2.97) | 10.03 (3.89)
  Measurement at 6 Months | 7.58 (3.53) | 9.84 (4.34)
Statistical Analysis 1: Comparison: Ablation Management vs Medical Management; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

8. Secondary Outcome: Improved Quality of Life Over 6 Months Compared to Baseline.
Description: The SF-36 questionnaire was administered to subjects at baseline, 1, 3 and 6 month visits. The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based Physical Component Score and Mental Component Score. The possible range for Physical Component Score and Mental Component Score is 0 to 100. The higher score, the better quality of life.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ablation Management | Medical Management
Number analyzed (Participants) | 138 | 72
Scores on a scale
  Physical Component Score at Baseline | 42.54 (10.45) | 42.26 (9.85)
  Physical Component Score at 1 Month | 45.61 (9.98) | 43.05 (10.46)
  Physical Component Score at 3 Months | 48.30 (9.76) | 43.99 (9.97)
  Physical Component Score at 6 Months | 49.12 (9.56) | 44.98 (9.59)
  Mental Component Score at Baseline | 47.19 (11.02) | 47.99 (12.13)
  Mental Component Score at 1 Month | 51.53 (10.34) | 48.96 (11.54)
  Mental Component Score at 3 Months | 53.42 (9.27) | 48.97 (10.52)
  Mental Component Score at 6 Months | 53.45 (9.07) | 50.06 (11.26)
Statistical Analysis 1: Comparison: Ablation Management vs Medical Management; Test type: Superiority or Other; p < 0.025, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the day of randomization to trial conclusion at the final 6 month follow-up. All adverse events were included even if the subject had a repeat procedure and the 6 month follow-up period was restarted.
Description: All adverse events (serious and nonserious) were recorded. Specific data about the event were entered into the electronic database. A planned hospital admission or unscheduled medical visit for atrial fibrillation that occurred within the follow-up period did not constitute an adverse event.
Arm/Group | Ablation Management | Medical Management
Serious Adverse Events (participants affected / at risk) | 41/138 | 3/72
Other Adverse Events (participants affected / at risk) | 25/138 | 3/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ablation Management (N=138) | Medical Management (N=72)
retroperitoneal bleed with right ureter obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0/0 (0)
heart failure (Cardiac disorders) | 2 (2) | 0/0 (0)
cardiac tamponade (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
pulmonary infiltrates (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
drop in hematocrit secondary to ablation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
anesthesia reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract infection with prolonged hospitalization (Renal and urinary disorders) | 1 (1) | 0 (0)
hypotension secondary to cardiac tamponade (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
hypotension/cardiogenic shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
pneumonia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
acute respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
stroke (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
post-procedure pericarditis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
pulmonary vein stenosis (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
pulmonary vein narrowing, symptomatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
chest pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
pericardial effusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
persistent atrial septal defect secondary to septal puncture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
gastrointestinal bleeds (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
AF with rapid ventricular response (Cardiac disorders) | 0 (0) | 1 (1)
coronary artery disease (Cardiac disorders) | 3 (3) | 0 (0)
bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
fever unknown origin with prolonged hospitalization (General disorders) | 1 (1) | 0 (0)
nausea and vomiting (General disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
congestive heart failure (Cardiac disorders) | 3 (3) | 0 (0)
sick sinus syndrome with pacemaker insertion (Cardiac disorders) | 1 (1) | 0 (0)
microcytic, hypochromic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Seriously elevated INR (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
mitral regurgitation with mitral valve replacement (Cardiac disorders) | 1 (1) | 0 (0)
chest discomfort secondary to mitral valve regurgitation (General disorders) | 1 (1) | 0 (0)
long QT with PVC's (Cardiac disorders) | 1 (1) | 0 (0)
rhythmol induced brugada effect (Cardiac disorders) | 1 (1) | 0 (0)
mitral regurgitation with surgical repair (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation Management (N=138) | Medical Management (N=72)
hematoma (Blood and lymphatic system disorders) | 16 (18) | 0 (0)
chest pain (General disorders) | 9 (10) | 0 (0)
bradycardia (Cardiac disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
- The study population was mostly Caucasian men.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No